CLINICAL TRIAL: NCT03932734
Title: Patient Satisfaction After Patient-specific Jawline Augmentation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veerle Van Mossevelde, Principal Investigator, Universitair Ziekenhuis Brussel
Other Study IDs: Survey Jawaug v1.0
Record Dates: First submitted 2019-04-15; First posted 2019-05-01 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Congenital Deformity of Face; Post-traumatic Deformity
Keywords: Satisfaction; Jawline augmentation; Transgender; Cosmetic jaw angle
MeSH Terms: conditions — Personal Satisfaction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- survey
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — Face-Q conversion table

SUMMARY:
The survey studies patient satisfaction after titanium patient specific jawline augmentation in congenital, post-trauma, deformity and transgender/cosmetic jaw angle/border deficiencies.

DETAILED DESCRIPTION:
Additively manufactured titanium implants have been pre-designed in the hospital department, further designed and manufactured by 2 Belgian companies. The issue is if all patients have satisfactory perception of the improvement of their morphology and the actual outcome of the procedure, and how theur social ineractions are perceived today.

ELIGIBILITY:
Inclusion Criteria:

- All lower jaw augmentation implants

Exclusion Criteria:

- N/A

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had lower jaw augmentation implants since 2014 not gender based
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Satisfaction/Quality of Life | 1 year
  By means of 4 surveys (social, psychological, outcome and satisfaction) based on FACE-Q. The scales can be used independently of the other scales.Higher scores reflect a better outcome. If missing data is less than 50% of the scale's items, insert the mean of the completed items. Use the Conversion Table to convert the raw summed scale score into a score from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Mommaerts, Prof Mult, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Vlaams Brabant, Belgium